CLINICAL TRIAL: NCT02608320
Title: A Randomized, Partially-blinded, Two-arm, Single-application, 3-way Crossover Study to Evaluate the Adherence of 2 Strengths of Newly Manufactured Samples and Aged Samples of a New Formulation (JNJ-35685-AAA-G016 and JNJ-35685-AAA-G021) of Fentanyl Transdermal System Compared With DURAGESIC Fentanyl Transdermal Patch in Healthy Subjects
Brief Title: A Study to Evaluate the Adherence of 2 Strengths of Newly Manufactured Samples and Aged Samples of a New Formulation (JNJ-35685-AAA-G016 and JNJ-35685-AAA-G021) of Fentanyl Transdermal System Compared With Duragesic Fentanyl Transdermal Patch in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Other
Other Study IDs: CR108060; FENPAI1025 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-11-17; First posted 2015-11-18 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Healthy; JNJ-35685-AAA-G016; JNJ-35685-AAA-G021; DURAGESIC; Fentanyl
MeSH Terms: interventions — Fentanyl; tyramine-deoxysorbitol

STUDY DESIGN:
Oversight: FDA-regulated Device: No

ARMS (24):
- Treatment Sequence (ACB) Position (RLR) (Experimental): Participants will receive treatment A (Duragesic 12.5 microgram per hour [mcg/h]) applied to right paraspinal side in period 1, then treatment C (aged JNJ- 35685-AAA-G016 12.5 mcg/h) applied to left paraspinal side in period 2 and then treatment B (New JNJ-35685- AAA-G016 12.5 mcg/h) applied to right paraspinal side in period 3.
  Interventions: Drug: Duragesic (Fentanyl Transdermal System [TDS] Small Patches); Drug: New JNJ-35685-AAA-G016 (Fentanyl TDS -Small Patches); Drug: Aged JNJ-35685-AAA-G016 (Fentanyl TDS Small Patches)
- Treatment Sequence (BAC) Position (RLR) (Experimental): Participants will receive treatment B applied to right paraspinal side in period 1, then treatment A applied to left paraspinal side in period 2 and then treatment C applied to right paraspinal side in period 3.
  Interventions: Drug: Duragesic (Fentanyl Transdermal System [TDS] Small Patches); Drug: New JNJ-35685-AAA-G016 (Fentanyl TDS -Small Patches); Drug: Aged JNJ-35685-AAA-G016 (Fentanyl TDS Small Patches)
- Treatment Sequence (CBA) Position (RLR) (Experimental): Participants will receive treatment C applied to right paraspinal side in period 1, then treatment B applied to left paraspinal side in period 2 and then treatment A applied to right paraspinal side in period 3.
  Interventions: Drug: Duragesic (Fentanyl Transdermal System [TDS] Small Patches); Drug: New JNJ-35685-AAA-G016 (Fentanyl TDS -Small Patches); Drug: Aged JNJ-35685-AAA-G016 (Fentanyl TDS Small Patches)
- Treatment Sequence (BCA) Position (RLR) (Experimental): Participants will receive treatment B applied to right paraspinal side in period 1, then treatment C applied to left paraspinal side in period 2 and then treatment A applied to right paraspinal side in period 3.
  Interventions: Drug: Duragesic (Fentanyl Transdermal System [TDS] Small Patches); Drug: New JNJ-35685-AAA-G016 (Fentanyl TDS -Small Patches); Drug: Aged JNJ-35685-AAA-G016 (Fentanyl TDS Small Patches)
- Treatment Sequence (CAB) Position (RLR) (Experimental): Participants will receive treatment C applied to right paraspinal side in period 1, then treatment A applied to left paraspinal side in period 2 and then treatment B applied to right paraspinal side in period 3.
  Interventions: Drug: Duragesic (Fentanyl Transdermal System [TDS] Small Patches); Drug: New JNJ-35685-AAA-G016 (Fentanyl TDS -Small Patches); Drug: Aged JNJ-35685-AAA-G016 (Fentanyl TDS Small Patches)
- Treatment Sequence (ABC) Position (RLR) (Experimental): Participants will receive treatment A applied to right paraspinal side in period 1, then treatment B applied to left paraspinal side in period 2 and then treatment C applied to right paraspinal side in period 3.
  Interventions: Drug: Duragesic (Fentanyl Transdermal System [TDS] Small Patches); Drug: New JNJ-35685-AAA-G016 (Fentanyl TDS -Small Patches); Drug: Aged JNJ-35685-AAA-G016 (Fentanyl TDS Small Patches)
- Treatment Sequence (ACB) Position (LRL) (Experimental): Participants will receive treatment A applied to left paraspinal side in period 1, then treatment C applied to right paraspinal side in period 2 and then treatment B applied to left paraspinal side in period 3.
  Interventions: Drug: Duragesic (Fentanyl Transdermal System [TDS] Small Patches); Drug: New JNJ-35685-AAA-G016 (Fentanyl TDS -Small Patches); Drug: Aged JNJ-35685-AAA-G016 (Fentanyl TDS Small Patches)
- Treatment Sequence (BAC) Position (LRL) (Experimental): Participants will receive treatment B applied to left paraspinal side in period 1, then treatment A applied to right paraspinal side in period 2 and then treatment C applied to left paraspinal side in period 3.
  Interventions: Drug: Duragesic (Fentanyl Transdermal System [TDS] Small Patches); Drug: New JNJ-35685-AAA-G016 (Fentanyl TDS -Small Patches); Drug: Aged JNJ-35685-AAA-G016 (Fentanyl TDS Small Patches)
- Treatment Sequence (CBA) Position (LRL) (Experimental): Participants will receive treatment C applied to left paraspinal side in period 1, then treatment B applied to right paraspinal side in period 2 and then treatment A applied to left paraspinal side in period 3.
  Interventions: Drug: Duragesic (Fentanyl Transdermal System [TDS] Small Patches); Drug: New JNJ-35685-AAA-G016 (Fentanyl TDS -Small Patches); Drug: Aged JNJ-35685-AAA-G016 (Fentanyl TDS Small Patches)
- Treatment Sequence (BCA) Position (LRL) (Experimental): Participants will receive treatment B applied to left paraspinal side in period 1, then treatment C applied to right paraspinal side in period 2 and then treatment A applied to left paraspinal side in period 3.
  Interventions: Drug: Duragesic (Fentanyl Transdermal System [TDS] Small Patches); Drug: New JNJ-35685-AAA-G016 (Fentanyl TDS -Small Patches); Drug: Aged JNJ-35685-AAA-G016 (Fentanyl TDS Small Patches)
- Treatment Sequence (CAB) Position (LRL) (Experimental): Participants will receive treatment C applied to left paraspinal side in period 1, then treatment A applied to right paraspinal side in period 2 and then treatment B applied to left paraspinal side in period 3.
  Interventions: Drug: Duragesic (Fentanyl Transdermal System [TDS] Small Patches); Drug: New JNJ-35685-AAA-G016 (Fentanyl TDS -Small Patches); Drug: Aged JNJ-35685-AAA-G016 (Fentanyl TDS Small Patches)
- Treatment Sequence (ABC) Position (LRL) (Experimental): Participants will receive treatment A applied to left paraspinal side in period 1, then treatment B applied to right paraspinal side in period 2 and then treatment C applied to left paraspinal side in period 3.
  Interventions: Drug: Duragesic (Fentanyl Transdermal System [TDS] Small Patches); Drug: New JNJ-35685-AAA-G016 (Fentanyl TDS -Small Patches); Drug: Aged JNJ-35685-AAA-G016 (Fentanyl TDS Small Patches)
- Treatment Sequence (DFE) Position (RLR) (Experimental): Participants will receive treatment D (Duragesic 100 mcg/h) applied to right paraspinal side in period 1, then treatment F (aged JNJ-35685-AAA-G021 100 mcg/h) applied to left paraspinal side in period 2 and then treatment E (new JNJ-35685-AAA-G021 100 mcg/h) applied to right paraspinal side in period 3.
  Interventions: Drug: Duragesic (Fentanyl TDS Large Patches); Drug: New JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches); Drug: Aged JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches)
- Treatment Sequence (EDF) Position (RLR) (Experimental): Participants will receive treatment E applied to right paraspinal side in period 1, then treatment D applied to left paraspinal side in period 2 and then treatment F applied to right paraspinal side in period 3.
  Interventions: Drug: Duragesic (Fentanyl TDS Large Patches); Drug: New JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches); Drug: Aged JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches)
- Treatment Sequence (FED) Position (RLR) (Experimental): Participants will receive treatment F applied to right paraspinal side in period 1, then treatment E applied to left paraspinal side in period 2 and then treatment D applied to right paraspinal side in period 3.
  Interventions: Drug: Duragesic (Fentanyl TDS Large Patches); Drug: New JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches); Drug: Aged JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches)
- Treatment Sequence (EFD) Position (RLR) (Experimental): Participants will receive treatment E applied to right paraspinal side in period 1, then treatment F applied to left paraspinal side in period 2 and then treatment D applied to right paraspinal side in period 3.
  Interventions: Drug: Duragesic (Fentanyl TDS Large Patches); Drug: New JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches); Drug: Aged JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches)
- Treatment Sequence (FDE) Position (RLR) (Experimental): Participants will receive treatment F applied to right paraspinal side in period 1, then treatment D applied to left paraspinal side in period 2 and then treatment E applied to right paraspinal side in period 3.
  Interventions: Drug: Duragesic (Fentanyl TDS Large Patches); Drug: New JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches); Drug: Aged JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches)
- Treatment Sequence (DEF) Position (RLR) (Experimental): Participants will receive treatment D applied to right paraspinal side in period 1, then treatment E applied to left paraspinal side in period 2 and then treatment F applied to right paraspinal side in period 3.
  Interventions: Drug: Duragesic (Fentanyl TDS Large Patches); Drug: New JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches); Drug: Aged JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches)
- Treatment Sequence (DFE) Position (LRL) (Experimental): Participants will receive treatment D applied to left paraspinal side in period 1, then treatment F applied to right paraspinal side in period 2 and then treatment E applied to left paraspinal side in period 3.
  Interventions: Drug: Duragesic (Fentanyl TDS Large Patches); Drug: New JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches); Drug: Aged JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches)
- Treatment Sequence (EDF) Position (LRL) (Experimental): Participants will receive treatment E applied to left paraspinal side in period 1, then treatment D applied to right paraspinal side in period 2 and then treatment F applied to left paraspinal side in period 3.
  Interventions: Drug: Duragesic (Fentanyl TDS Large Patches); Drug: New JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches); Drug: Aged JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches)
- Treatment Sequence (FED) Position (LRL) (Experimental): Participants will receive treatment F applied to left paraspinal side in period 1, then treatment E applied to right paraspinal side in period 2 and then treatment D applied to left paraspinal side in period 3.
  Interventions: Drug: Duragesic (Fentanyl TDS Large Patches); Drug: New JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches); Drug: Aged JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches)
- Treatment Sequence (EFD) Position (LRL) (Experimental): Participants will receive treatment E applied to left paraspinal side in period 1, then treatment F applied to right paraspinal side in period 2 and then treatment D applied to left paraspinal side in period 3.
  Interventions: Drug: Duragesic (Fentanyl TDS Large Patches); Drug: New JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches); Drug: Aged JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches)
- Treatment Sequence (FDE) Position (LRL) (Experimental): Participants will receive treatment F applied to left paraspinal side in period 1, then treatment D applied to right paraspinal side in period 2 and then treatment E applied to left paraspinal side in period 3.
  Interventions: Drug: Duragesic (Fentanyl TDS Large Patches); Drug: New JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches); Drug: Aged JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches)
- Treatment Sequence (DEF) Position (LRL) (Experimental): Participants will receive treatment D applied to left paraspinal side in period 1, then treatment E applied to right paraspinal side in period 2 and then treatment F applied to left paraspinal side in period 3.
  Interventions: Drug: Duragesic (Fentanyl TDS Large Patches); Drug: New JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches); Drug: Aged JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches)

INTERVENTIONS:
Drug: Duragesic (Fentanyl Transdermal System [TDS] Small Patches) — Duragesic 12.5 mcg/h (Treatment A) in either period 1, 2 or 3 as per treatment sequence, applied to the paraspinal region of the back for 72 hours.
  Arms: Treatment Sequence (ABC) Position (LRL); Treatment Sequence (ABC) Position (RLR); Treatment Sequence (ACB) Position (LRL); Treatment Sequence (ACB) Position (RLR); Treatment Sequence (BAC) Position (LRL); Treatment Sequence (BAC) Position (RLR); Treatment Sequence (BCA) Position (LRL); Treatment Sequence (BCA) Position (RLR); Treatment Sequence (CAB) Position (LRL); Treatment Sequence (CAB) Position (RLR); Treatment Sequence (CBA) Position (LRL); Treatment Sequence (CBA) Position (RLR)
Drug: New JNJ-35685-AAA-G016 (Fentanyl TDS -Small Patches) — New JNJ-35685-AAA-G016 12.5 mcg/h (Treatment B) in either period 1, 2 or 3 as per treatment sequence, applied to the paraspinal region of the back for 72 hours.
  Arms: Treatment Sequence (ABC) Position (LRL); Treatment Sequence (ABC) Position (RLR); Treatment Sequence (ACB) Position (LRL); Treatment Sequence (ACB) Position (RLR); Treatment Sequence (BAC) Position (LRL); Treatment Sequence (BAC) Position (RLR); Treatment Sequence (BCA) Position (LRL); Treatment Sequence (BCA) Position (RLR); Treatment Sequence (CAB) Position (LRL); Treatment Sequence (CAB) Position (RLR); Treatment Sequence (CBA) Position (LRL); Treatment Sequence (CBA) Position (RLR)
Drug: Aged JNJ-35685-AAA-G016 (Fentanyl TDS Small Patches) — Aged JNJ-35685-AAA-G016 12.5 mcg/h (Treatment C) in either period 1, 2 or 3 as per treatment sequence, applied to the paraspinal region of the back for 72 hours.
  Arms: Treatment Sequence (ABC) Position (LRL); Treatment Sequence (ABC) Position (RLR); Treatment Sequence (ACB) Position (LRL); Treatment Sequence (ACB) Position (RLR); Treatment Sequence (BAC) Position (LRL); Treatment Sequence (BAC) Position (RLR); Treatment Sequence (BCA) Position (LRL); Treatment Sequence (BCA) Position (RLR); Treatment Sequence (CAB) Position (LRL); Treatment Sequence (CAB) Position (RLR); Treatment Sequence (CBA) Position (LRL); Treatment Sequence (CBA) Position (RLR)
Drug: Duragesic (Fentanyl TDS Large Patches) — Duragesic 100 mcg/h (Treatment D) in either period 1, 2 or 3 as per treatment sequence, applied to the paraspinal region of the back for 72 hours, applied to the paraspinal region of the back for 72 hours.
  Arms: Treatment Sequence (DEF) Position (LRL); Treatment Sequence (DEF) Position (RLR); Treatment Sequence (DFE) Position (LRL); Treatment Sequence (DFE) Position (RLR); Treatment Sequence (EDF) Position (LRL); Treatment Sequence (EDF) Position (RLR); Treatment Sequence (EFD) Position (LRL); Treatment Sequence (EFD) Position (RLR); Treatment Sequence (FDE) Position (LRL); Treatment Sequence (FDE) Position (RLR); Treatment Sequence (FED) Position (LRL); Treatment Sequence (FED) Position (RLR)
Drug: New JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches) — New JNJ-35685-AAA-G021 100 mcg/h (Treatment E) in either period 1, 2 or 3 as per treatment sequence, applied to the paraspinal region of the back for 72 hours.
  Arms: Treatment Sequence (DEF) Position (LRL); Treatment Sequence (DEF) Position (RLR); Treatment Sequence (DFE) Position (LRL); Treatment Sequence (DFE) Position (RLR); Treatment Sequence (EDF) Position (LRL); Treatment Sequence (EDF) Position (RLR); Treatment Sequence (EFD) Position (LRL); Treatment Sequence (EFD) Position (RLR); Treatment Sequence (FDE) Position (LRL); Treatment Sequence (FDE) Position (RLR); Treatment Sequence (FED) Position (LRL); Treatment Sequence (FED) Position (RLR)
Drug: Aged JNJ-35685-AAA-G021 (Fentanyl TDS Large Patches) — Aged JNJ-35685-AAA-G021 100 mcg/h (Treatment F) in either period 1, 2 or 3 as per treatment sequence, applied to the paraspinal region of the back for 72 hours.
  Arms: Treatment Sequence (DEF) Position (LRL); Treatment Sequence (DEF) Position (RLR); Treatment Sequence (DFE) Position (LRL); Treatment Sequence (DFE) Position (RLR); Treatment Sequence (EDF) Position (LRL); Treatment Sequence (EDF) Position (RLR); Treatment Sequence (EFD) Position (LRL); Treatment Sequence (EFD) Position (RLR); Treatment Sequence (FDE) Position (LRL); Treatment Sequence (FDE) Position (RLR); Treatment Sequence (FED) Position (LRL); Treatment Sequence (FED) Position (RLR)

SUMMARY:
The purpose of this study is to evaluate the cumulative adhesion percentage for the test products and the reference products for both small and large patches.

DETAILED DESCRIPTION:
This is a randomized (study medication assigned to participants by chance), single-center, parallel-group single-application, modified 3-way crossover study. Each participant will receive the marketed reference formulation (DURAGESIC) or the JNJ-35685-AAA-G016 or JNJ-35685-AAA-G021 fentanyl transdermal system (TDS). The study consists of a screening phase within 21 and 2 days before the first TDS application of the first period; a partially-blinded treatment phase consisting of 3 single-application treatment periods; and end-of-study or withdrawal assessments done upon completion of the 72-hour adhesion assessment on Day 5 of Period 3 or upon withdrawal. A 7- to 16-day washout period will separate the treatment periods, commencing at transdermal patch removal. The duration of participation in the study for an individual participant will be 31 days to a maximum of 68 days (including screening and follow-up visits). Participants will be primarily evaluated for cumulative adhesion percentage. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening. This determination must be recorded in the participant's source documents and initialed by the investigator
* A woman of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) test at screening and urine pregnancy test at Day -1 of the first treatment period
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control example, either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 3 months after completion of the study
* Participant must be willing and able to adhere to the prohibitions and restrictions specified in this protocol
* Body mass index (BMI) between 18 and 30 kilogram per square meter (kg/m^2), inclusive, and a body weight of not less than 50 kg

Exclusion Criteria:

* Participant has a history of or current clinically significant medical illness including but not limited to, cardiac arrhythmias or other cardiac disease; hematologic disease; coagulation disorders (including any abnormal bleeding or blood dyscrasias); lipid abnormalities; significant pulmonary disease, including bronchospastic respiratory disease; diabetes mellitus; hepatic or renal insufficiency (creatinine clearance below 60 milliliter per minute [mL/min]); thyroid disease; neurologic or psychiatric disease; infection; or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening as deemed appropriate by the investigator
* Clinically significant abnormal physical examination, vital signs or 12 lead ECG at screening as deemed appropriate by the investigator
* Use of medications or treatments that would significantly influence or exaggerate patch adhesion or that would alter inflammatory or immune response to the study product (example antihistamines, systemic or topical corticosteroids, cyclosporine, tacrolimus, cytotoxic drugs, immune globulin, Bacillus Calmette-Guerin (BCG), monoclonal antibodies, radiation therapy)
* History of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (4th edition) criteria within 5 years before screening or positive test result(s) for alcohol and/or drugs of abuse (such as barbiturates, opiates, cocaine, cannabinoids, amphetamines, and benzodiazepines) at screening. Participants must not use tobacco products, including all nicotine use, example, cigarettes, cigars, chewing tobacco, patch, gum

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-11-17 (Actual); Primary Completion 2016-04-13 (Actual); Study Completion 2016-04-13 (Actual)

PRIMARY OUTCOMES:
Cumulative Adhesion Percentage | Time of patch application up to patch removal (up to 72 hours)
  The actual percentages of patch adhesion will be estimated according to the Food and Drug Administration (FDA) 0-4 scoring system. An estimated percentage of adhesion, to a whole integer, will be obtained (FDA 0-4 [%] scoring) where 0=greater than or equal to (>=) 90% adhered (essentially no lift off the skin); 1= >= 75% to < 90% adhered (some edges only lifting off the skin); 2 = ≥ 50% to < 75% adhered (less than half of the patch lifting off the skin); 3 = > 0% to < 50% adhered but not detached (more than half of the patch lifting off the skin without falling off); 4 = 0% adhered - patch detached (patch completely off the skin).

SECONDARY OUTCOMES:
Time to First Unacceptable Score | 12, 24, 36, 48, 60, and 72 hour following patch application
  Time to first unacceptable score that is < 75% adhered will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Cypress, California, United States